CLINICAL TRIAL: NCT05547815
Title: Single Arm, Single Center Phase IV Clinical Trial to Evaluate the Immune Persistence and Safety of Freeze-dried Human Rabies Vaccine (Vero Cell)
Brief Title: Observation on the Immune Persistence of People Aged 10-60 Years Old Immunized With Five Doses of Rabies Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changchun Zhuoyi Biological Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZY201909001
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Rabies; Antibody
Keywords: rabies vaccine; antibody; persistence
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental): 5 doses of rabies vaccine
  Interventions: Biological: 5 doses program

INTERVENTIONS:
Biological: 5 doses program — Inoculate 5 doses of rabies vaccine, and collect blood at fixed time points to detect neutralizing antibody

SUMMARY:
Evaluation of immune persistence after rabies vaccination in 150 people.

DETAILED DESCRIPTION:
150 subjects aged 10-60 were recruited to inoculate the frozen human rabies vaccine (Vero cells) produced and marketed by Changchun Zhuoyi Biological Co., Ltd. in the whole process of 0, 3, 7, 14 and 28 day immunization. The immunogenicity persistence and safety of the test vaccine were evaluated 14 days, 6 months and 12 months after the whole process of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 10-60 years old；
* Temperature on the day of admission≤37.0 ° C (axillary temperature).

Exclusion Criteria:

* Have a history of rabies vaccine immunization or use of rabies virus passive immunization agents；
* Has been diagnosed with congenital or acquired immunodeficiency disease;
* Pregnancy (including positive urine pregnancy test) or lactation, planned pregnancy preparation within 2 months.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 149 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
positive conversion rate evaluation (6 months) | 6 months
  Evaluate the positive conversion rate 6 months after vaccination of rabies vaccine according to the 5-dose immunization program
antibody titer evaluation (6 months) | 6 months
  Evaluate the antibody titer of serum neutralizing antibody 6 months after vaccination of rabies vaccine according to the 5-dose immunization program
positive conversion rate evaluation (12 months) | 12 months
  Evaluate the positive conversion rate 12 months after vaccination of rabies vaccine according to the 5-dose immunization program
antibody titer evaluation (12 months) | 12 months
  Evaluate the antibody titer of serum neutralizing antibody 12 months after vaccination of rabies vaccine according to the 5-dose immunization program

CONTACTS AND LOCATIONS:
Overall Officials: Li Miao, Dr, Study Director — Changchun Zhuoyi Biological Co., Ltd
Locations (1):
- Changchun Zhuoyi Biological Co., Ltd, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
all data of antibody titer .
Supporting Information: Study Protocol, CSR
Time Frame: before December 2022.
Access Criteria: public for all.